CLINICAL TRIAL: NCT04292834
Title: A Registered Cohort Study of Immune-Mediated Neuropathies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ning Wang, MD., PhD., Director, First Affiliated Hospital of Fujian Medical University
Other Study IDs: MRCTA，ECFAH of FMU2019217
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will provide further insights into the natural course of the disease about Immune-Mediated Neuropathies including clinical features，progression, related antibody spectrum and drug treatment effect.

ELIGIBILITY:
Inclusion Criteria:

- 1. Outpatient or inpatient 2. Meet the diagnostic criteria of various inflammatory peripheral neuropathy. 3. Voluntary participation and informed consent signed by the applicant or his/her family.

4. Age 18 or above

Exclusion Criteria:

1. Severe complications
2. Poor prognosis (<1 year survival)
3. Severe mental disorder and inability to cooperate with the examination.
4. Age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with GBS,CIDP,MMN who are diagnosied in the First Affiliated Hospital of Fujian Medical Universtiy and Beijing Tiantan Hospital, Capital Medical University by two neurolgists
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-29 (Actual); Primary Completion 2022-01-19 (Estimated); Study Completion 2025-01-19 (Estimated)

PRIMARY OUTCOMES:
The correlation between clinical phenotypes and Serum antibodies | from date of enrollment until the date of death from any cause,assessed up to 20 years
  Different clinical subtypes of GBS and CIDP have different course and prognosis.It may be related to different serum antibodies.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Department of Neurology,First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian

IPD SHARING:
Plan to Share IPD: No